CLINICAL TRIAL: NCT00448448
Title: Bracing in Adolescent Idiopathic Scoliosis Trial (BrAIST)
Acronym: BrAIST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped for efficacy
Sponsor: Stuart L. Weinstein, MD (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Shriners Hospitals for Children (Other); Children's Mercy Hospital Kansas City (Other); University of Rochester (Other)
Responsible Party: Sponsor-Investigator, Stuart L. Weinstein, MD, Professor of Orthopaedics and Rehabilitation, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200108052; R01AR052113 (NIH)
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2019-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; orthotics; bracing; partially randomized preference design
MeSH Terms: interventions — Braces; Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor(s) are blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brace (Active Comparator): This study involves full-time, rigid TLSO's only. Braced subjects are followed every six months with radiography, clinical exam and self-reported evaluations of health and functioning. Orthotic evaluations are conducted every 6 months as as necessary to maintain brace fit and function.
  Interventions: Device: Brace
- Observation (Active Comparator): Observation. Observed subjects are followed every six months with radiography, clinical exam and self-reported evaluations of health and functioning.
  Interventions: Other: Observation

INTERVENTIONS:
Device: Brace — Brace (TLSO) applied for at least 18 hours per day. Wear time measured using a temperature monitor. Clinical, radiographic, and self-report follow-up every 6 months.
  Arms: Brace
Other: Observation — Clinical, radiographic, and self-report follow-up every 6 months.
  Arms: Observation

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a structural curve of the spine with no clear underlying cause. Bracing is currently the standard of care for preventing curve progression and treating AIS. However, the effectiveness of bracing remains unclear. The purpose of this study is to compare the risk of curve progression in adolescents with AIS who wear a brace versus those who do not and to determine whether there are reliable factors that can predict the usefulness of bracing for a particular individual with AIS.

DETAILED DESCRIPTION:
AIS is characterized by a lateral curvature of the spine greater than 10 degrees plus rotation of the spinal vertebrae. AIS is found in adolescents between the age of 10 and time of skeletal maturity. Progression of a spinal curve to 50 degrees suggests a high risk for continued curve progression throughout adulthood and usually indicates the need for spinal fusion surgery. Only about 10 percent of adolescents with AIS end up having curves that progress and require surgical intervention. While certain risk factors for curve progression have been identified, there is no reliable way of estimating the likelihood of needing surgery. Bracing is currently the standard of care for treating AIS. However, the effectiveness of bracing remains unclear, and it is unknown which adolescents in particular may benefit from bracing. Therefore, adolescents undergo bracing without knowing their likelihood of avoiding surgery. The purpose of this study is to compare the risk of curve progression in adolescents with AIS who wear a brace versus those who do not and to determine whether there are reliable factors that can predict the usefulness of bracing for a particular individual with AIS. The study will also evaluate the best dosing and duration schedule and how bracing affects quality of life, functioning, and psychosocial adjustment among participants.

Participation in this study will last until a participant reaches skeletal maturity or their spinal curve progresses to 50 degrees, after which usual care will continue. Participants will either be 1)randomly assigned to a treatment or 2) may decline randomization and choose their own treatment arm. Study visits will occur every 6 months at an orthopaedic surgeon's office and will include x-rays, a clinical exam, and questionnaires. Participants assigned to braces will be instructed to wear the brace at least 18 hours per day. Temperature monitors placed in the brace will be used to determine the actual wear time by each participant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS
* Skeletally immature (Risser grade 0, 1, or 2)
* Pre-menarchal or post-menarchal by no more than 1 year
* Primary Cobb angle between 20 and 40 degrees
* Curve apex caudal to T7 vertebrae
* Physical and mental ability to adhere to bracing protocol
* Ability to read and understand English, Spanish, or French
* Documented insurance coverage and/or personal willingness to pay for treatment

Exclusion Criteria:

* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical or orthotic treatment for AIS

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 383 (Actual)
Dates: Start 2007-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L. Weinstein, MD, Principal Investigator — University of Iowa; Lori A. Dolan, PhD, Study Director — University of Iowa
Locations (25):
- United States (22):
  - Children's Hospital Central California, Madera, California
  - Shriners Hospital of Northern California, Sacramento, California
  - Rady Childrens Hospital, San Diego, California
  - Alfred I. duPont Hospital for Children and Nemours Children's Clinic, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Shriner's Hospital for Children, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Shriners Hospitals for Children - Lexington, Lexington, Kentucky
  - Children's Hospital Boston, Boston, Massachusetts
  - Shriners Hospitals for Children - Minneapolis, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics., Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Shriners Hospitals for Children - St. Louis, St Louis, Missouri
  - Carrie Tingley Hospital, Albuquerque, New Mexico
  - Hospital for Special Surgery, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Shriners Hospitals for Children - Salt Lake City, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- Canada (3):
  - BC Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - Shriner's Hospital for Children, Montreal, Quebec

REFERENCES:
- [Background] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Design of the Bracing in Adolescent Idiopathic Scoliosis Trial (BrAIST). Spine (Phila Pa 1976). 2013 Oct 1;38(21):1832-41. doi: 10.1097/01.brs.0000435048.23726.3e. PMID 24026162
- [Result] Schwieger T, Campo S, Weinstein SL, Dolan LA, Ashida S, Steuber KR. Body Image and Quality-of-Life in Untreated Versus Brace-Treated Females With Adolescent Idiopathic Scoliosis. Spine (Phila Pa 1976). 2016 Feb;41(4):311-9. doi: 10.1097/BRS.0000000000001210. PMID 26555827
- [Result] Dolan LA, Donzelli S, Zaina F, Weinstein SL, Negrini S. Adolescent Idiopathic Scoliosis Bracing Success Is Influenced by Time in Brace: Comparative Effectiveness Analysis of BrAIST and ISICO Cohorts. Spine (Phila Pa 1976). 2020 Sep 1;45(17):1193-1199. doi: 10.1097/BRS.0000000000003506. PMID 32205704
- [Result] Dolan LA, Weinstein SL, Dobbs MB, Flynn JMJ, Green DW, Halsey MF, Hresko MT, Krengel WF 3rd, Mehlman CT, Milbrandt TA, Newton PO, Price N, Sanders JO, Schmitz ML, Schwend RM, Shah SA, Song K, Talwalkar V. BrAIST-Calc: Prediction of Individualized Benefit From Bracing for Adolescent Idiopathic Scoliosis. Spine (Phila Pa 1976). 2024 Feb 1;49(3):147-156. doi: 10.1097/BRS.0000000000004879. Epub 2023 Nov 23. PMID 37994691
- [Result] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17;369(16):1512-21. doi: 10.1056/NEJMoa1307337. Epub 2013 Sep 19. PMID 24047455
- [Result] Schwieger T, Campo S, Weinstein SL, Dolan LA, Ashida S, Steuber KR. Body Image and Quality of Life and Brace Wear Adherence in Females With Adolescent Idiopathic Scoliosis. J Pediatr Orthop. 2017 Dec;37(8):e519-e523. doi: 10.1097/BPO.0000000000000734. PMID 26886460
- See also: BrAIST-Calc is an online aid for patients with Adolescent Idiopathic Scoliosis who want to estimate their personal risk of scoliosis surgery with and without bracing treatment. — http://braistcalc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 25 centers in the US and Canada (see list of participating centers). The first subject was enrolled in April 2007 and the last in February 2011.
Period: Overall Study
Arm/Group | Brace | Observation
Started | 246 | 137
Completed | 146 | 96
Not Completed | 100 | 41
Not completed — Withdrawal by Subject | 13 | 2
Not completed — On protocol when study ended | 83 | 36
Not completed — Lost to Follow-up | 2 | 1
Not completed — Wrong diagnosis (n=3) or other | 2 | 1
Not completed — Signed consent lost | 0 | 1

BASELINE CHARACTERISTICS:
Population: Age, gender, race, height, Scoliosis Research Society curve classification, Cobb angle, Risser grade
Groups:
- Brace: This study involves full-time, rigid TLSO's only. Braced subjects are followed every six months with radiography, clinical exam and self-reported evaluations of health and functioning.
  Brace: Brace (TLSO) prescribed for at least 18 hours per day. Wear time measured using a temperature monitor. Orthotic evaluations are conducted every 6 months and as necessary to maintain brace fit and function.
- Total: Total of all reporting groups
Arm/Group | Brace | Observation | Total
Number analyzed (Participants) | 146 | 96 | 484
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 146 | 96 | 242
  (all) | 12.7 (1.0) | 12.7 (1.2) | 12.7 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 146 | 96 | 242
  Female | 135 | 86 | 221
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  number analyzed (Participants) | 146 | 96 | 242
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 11 | 11 | 22
  White | 116 | 73 | 189
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 3 | 14
Risser grade [Number; unit: participants] — The Risser grade is a measure of the amount of ossification and eventual fusion of the iliac apophysis reflecting skeletal maturity. Grades range from 0 to 5, with higher grades indicating greater maturity. Patients who are classified as being Risser 0, 1 or 2 are regarded as having significant skeletal growth remaining and therefore as being at higher risk for scoliosis progression relative to those classified as Risser 3 or greater. Girls are generally considered skeletally mature at Risser 4 or greater; boys at Risser 5.
  participants
    0: number analyzed (Participants) | 146 | 96 | 242
    0 | 82 | 60 | 142
    1: number analyzed (Participants) | 146 | 96 | 242
    1 | 45 | 19 | 64
    2: number analyzed (Participants) | 146 | 96 | 242
    2 | 15 | 12 | 27
    3: number analyzed (Participants) | 146 | 96 | 242
    3 | 2 | 3 | 5
    4: number analyzed (Participants) | 146 | 96 | 242
    4 | 1 | 0 | 1
    5: number analyzed (Participants) | 146 | 96 | 242
    5 | 1 | 0 | 1
    MISSING: number analyzed (Participants) | 146 | 96 | 242
    MISSING | 0 | 2 | 2
Cobb angle [Mean (Standard Deviation); unit: angle in degrees] — The Cobb angle is the most frequently used measurement of the magnitude of the curvature of the spine, and is a function of the tilt of the vertebrae at the top and bottom of the spinal curvature. A Cobb angle of 10 degrees or greater in association with rotation of the vertebrae indicates the presence of scoliosis.
  angle in degrees
    number analyzed (Participants) | 146 | 96 | 242
    (all) | 30.5 (5.8) | 30.3 (6.5) | 30.4 (6.0)
Curve type using SRS classification [Number; unit: participants] — The Scoliosis Research Society has classified scoliosis according to the apex of the curvature(s).
  participants
    Thoracic: number analyzed (Participants) | 146 | 96 | 242
    Thoracic | 38 | 21 | 59
    Thoracolumbar: number analyzed (Participants) | 146 | 96 | 242
    Thoracolumbar | 19 | 13 | 32
    Lumbar: number analyzed (Participants) | 146 | 96 | 242
    Lumbar | 5 | 4 | 9
    Double Major: number analyzed (Participants) | 146 | 96 | 242
    Double Major | 37 | 32 | 69
    Double Thoracic: number analyzed (Participants) | 146 | 96 | 242
    Double Thoracic | 15 | 7 | 22
    Thoracic/Thoracolumbar: number analyzed (Participants) | 146 | 96 | 242
    Thoracic/Thoracolumbar | 20 | 13 | 33
    Triple: number analyzed (Participants) | 146 | 96 | 242
    Triple | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Maturity With a Cobb Angle of <50 Degrees (Successful Outcome)
Time Frame: Skeletal maturity and the Cobb angle were measured at baseline and at each 6-month follow-up. Subjects were followed until they reached criteria for either success or failure. The average duration of follow-up was 23.67 months.
Population: The primary analysis included all patients who had completed the trial by January 2013, including 116 patients from the randomized arm and 126 from the preference arm.
Measure: Number; unit: percentage of patient successes
Arm/Group | Brace | Observation
Number analyzed (Participants) | 146 | 96
percentage of patient successes | 72 | 48
Statistical Analysis 1: Comparison: Brace vs Observation; Test type: Superiority or Other; p < 0.0267, Regression, Logistic; The success rate was adjusted for the propensity score (probability of receiving a brace) and the duration of follow-up; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.08 to 3.46]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected continuously while subjects were on protocol, which was an average of 23.67 months
Description: Multiple events per participant were recorded
Arm/Group | Brace | Observation
Serious Adverse Events (participants affected / at risk) | 1/146 | 0/96
Other Adverse Events (participants affected / at risk) | 71/146 | 36/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brace (N=146) | Observation (N=96)
Anxiety and Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Subject was hospitalized for anxiety and depression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brace (N=146) | Observation (N=96)
SnoMed term not found (Reproductive system and breast disorders) | 0 (0) | 1 (1) — non-specific report of abnormal breast development
Arm Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Backache (Musculoskeletal and connective tissue disorders) | 30 (37) | 25 (29)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Dislocation of patellofemoral joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eruption of skin (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) — Rash
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fracture of great toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headaches (Nervous system disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Numbness of limb (Nervous system disorders) | 4 (5) | 2 (2) — Report of either or both arm and leg numbness and/or tingling
Numbness of saddle area (Nervous system disorders) | 1 (1) | 0 (0) — Report of numbness in hip area
Pain (Nervous system disorders) | 1 (1) | 0 (0) — Report of side pain
Shoulder pain (Nervous system disorders) | 5 (5) | 2 (2)
Suicidal thoughts (Psychiatric disorders) | 1 (1) | 0 (0) — Subject with history of depression; event not related to protocol
Superficial bruising (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Superficial ulcer of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Vaso vagal episode (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Report of asthma exacerbation
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee reflex abnormal (Nervous system disorders) | 1 (1) | 0 (0) — Report of asymmetrical patella reflexes
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early due to efficacy. 119 subjects were still on protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No